CLINICAL TRIAL: NCT03057678
Title: Evaluating the Pre-Positioning Frame for Robotic Acoustic Neuroma Removal Surgery
Acronym: PPF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants have been enrolled. The PI Is leaving the institution and we wish to close the study at this time.
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Robert F. Labadie, Vice Chair, Chief Research Officer, Professor of Otolaryngology-Head and Neck Surgery, Professor of Biomedical Engineering, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 151347; R01DC012593 (NIH)
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Acoustic Neuroma
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Testing of Pre-Positioning Frame (Experimental): Placement of bone screws, CT scanning, Surgical planning, Robot motion planning
  Interventions: Other: Testing of Pre-Positioning Frame

INTERVENTIONS:
Other: Testing of Pre-Positioning Frame — Placement of bone screws, CT scanning, Surgical planning, Robot motion planning

SUMMARY:
Otologic surgery often involves a mastoidectomy to safely access the inner ear. In this procedure, a portion of the mastoid part of the temporal bone is removed. The surgery is lengthy and challenging because many critical structures are embedded in the mastoid and are difficult to identify and accurately remove with a surgical drill. In previous work, the investigators developed a compact, bone-attached robot to automate mastoidectomy drilling for translabyrinthine acoustic neuroma removal (TANR). The robot does not attach directly to the bone. Instead, a rigid surgical fixture which the investigators call a prepositioning frame (PPF) is attached to the temporal bone, and the robot attaches to the PPF. Attaching the robot to the participant eliminates the need for an expensive image guidance system to compensate for participant motion, but requires a compact robot with a limited range of motion. The PPF supports the robot on the head such that a planned mastoidectomy volume is within the robot's range of motion. In this study, the investigators plan to test the PPF by attaching it to ten participants. By processing an intraoperative CT scan of the attached PPF, the investigators will measure the percentage of each planned mastoidectomy that would be reachable if the robot were attached. The investigators will also measure the time required to attach the PPF. The data the investigators acquire will enable further improvements to the PPF design, which would be advantageous before proceeding to robotic drilling experiments.

DETAILED DESCRIPTION:
Mastoidectomy is a common otologic surgical procedure in which all or part of the mastoid portion of the temporal bone is removed with a surgical drill. The procedure is performed to treat diseases and infections such as mastoiditis and cholesteatoma, and is also performed as one step of other surgeries, such as the facial recess approach for cochlear implantation (CI) or the translabyrinthine approach for acoustic neuroma removal (TANR). The investigators are working on a new medical device to assist specifically with the TANR procedure. The focus of this study is one component of this device, the pre-positioning frame (PPF).

TANR surgery is performed to remove benign tumors on the auditory nerve which can cause severe hearing and balance problems if not removed. The current standard of care is a mastoidectomy, followed by a labyrinthectomy (excision of the labyrinth of the inner ear) to gain access to the skull base, specifically the internal auditory canal (IAC), where tumors are located.

Several critical anatomical structures are embedded in the mastoid bone, including the facial nerve, which controls motion of the face, large blood vessels such as the carotid artery and intracranial continuation of the jugular vein, and the tegmen, which is the boundary between the mastoid and the brain. Surgeons are specially trained to recognize and avoid these structures when drilling. Drilling for TANR surgery often takes several hours due to slow advancement of the drill through hard bone in the labyrinth region. After this drilling is when the most delicate and critical portion of the surgery begins i.e. removal of the acoustic neuroma. The investigators hypothesize that a robot, guided by pre-operative images, can perform the drilling for TANR surgery while preserving safe margins around the critical structures thus enabling surgeons to focus on the delicate, final stage of TANR surgery.

There are several robotic systems available for orthopedic drilling procedures such as joint arthroplasty and resurfacing. These systems include the RIO System (Stryker Mako, Ft. Lauderdale, FL, USA), the ROBODOC Surgical System (Think Surgical Corp., Fremont, CA, USA) and the CASPAR (URS Ortho GMBH & Co. KG, Rastatt, Germany). However, these systems have not been shown accurate enough to perform TANR surgery safely, and rely on expensive image guidance systems to continuously track the patient's position relative to the robot, in order to ensure that the robot-guided drill stays within safe margins.

The investigators previously designed a small light-weight robot that can be attached to the bone of a patient's head, and provide the required accuracy for TANR surgery without an expensive image guidance system.

To reach an entire mastoidectomy volume for TANR surgery, our robot must be correctly positioned relative to a patient's temporal bone anatomy. The investigators hypothesize that a rigid fixture, which the investigators call a pre-positioning frame (PPF), can correctly position our robot to complete drilling for TANR surgery on the patient population. The goal of this study is to investigate the first step in implementing this system by attaching a PPF to a patient who is undergoing a standard TANR surgery in order to better understand the time it takes to do this step and optimize the surgical workflow.

The PPF, attaches directly to the participants head behind the ear, using bone screws adapted from cranial reconstruction hardware. These bone screws are typically used in this area of the skull and placed at a similar penetration depth of 3.5 mm. The safety margin from tip of the screw to the inside skull surface will be 0.25mm In a future study, the robot would then attach to fiducial markers on the top surface of the PPF. Our current PPF design incorporates data from ten robotic drilling experiments. Six trials were performed on excised temporal bones, and four were performed on full cadaver heads. Using results from these experiments, the investigators improved the shape of the PPF to optimally reach the range of planned TANR mastoidectomy volumes, and also improved the legs of the PPF to facilitate rapid and secure implantation of bone screws.

The surgical workflow the investigators plan for a full robotic mastoidectomy will be described here for context, but to be clear, steps 7, 8, and 10 will not be performed in the proposed study.

1. Prior to surgery, a surgeon manually segments a mastoidectomy volume in a preoperative CT image using investigational software created for this purpose.
2. During surgery, the PPF is anchored to the temporal bone with self-drilling bone screws.
3. An intraoperative CT scan is acquired of the participants's head with the PPF attached using a portable CT scanner.
4. The intraoperative CT image is registered to the preoperative CT and the pre-operative segmentations are transformed to the intraoperative CT using the registration.
5. Fiducial markers on the PPF are localized in the intraoperative CT image, allowing the pre-operative segmentation data to be transformed to the intraoperative CT image space.
6. Robot motion is automatically planned using investigational mastoidectomy planning software.
7. (The robot is fastened to the fiducial markers on the PPF, and is activated to execute the drill trajectory. The surgeon retains supervisory control over the robot and can stop or alter its speed if necessary).
8. (The robot is removed from the PPF following completion of drilling).
9. The PPF is removed from the participant by loosening the bone screws.
10. (The surgeon completes the manual surgical actions that follow mastoidectomy drilling, such as removal of IAC tumors.) The investigators plan to clinically validate the improved PPF design by performing the steps above (excluding steps 7, 8, and 10) on ten participants. Note that the PPF will be removed directly after step 5 when the CT image has been registered. Using previously developed robotic mastoidectomy planning software (step 6), the investigators will calculate the percentage of each TANR mastoidectomy that is reachable for an attached PPF configuration. Step 6 will be done once the images have been collected and will not impact the clinical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients 21-80 years old undergoing TANR who consent to participation.
* Preop Head CT scan as part of routine care.
* Skull thickness a minimum of 3.75mm in planned attachment areas.

Exclusion Criteria:

* Pregnant women. As per standard of care in preparation for surgery, all females of childbearing age will undergo a pregnancy test during the medical evaluation for surgery.
* Patients with severe comorbidities, such as chronic otitis media, history of stroke, brain trauma, or hydrocephalus.
* Patients with a history of allergic reactions to lidocaine.
* Patients with severe anatomical abnormality of the temporal bone.
* Patients with history of allergic reaction to titanium, because the bone screws used in this study are made of a titanium alloy.
* Patients who are at unacceptable risk for general anesthesia.
* Patients who are at unacceptable risk for the intraoperative CT scan(s).
* Patients who are unable to give informed consent.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Time in minutes required to attach the PPF. | From PPF anchored to temporal bone until bone screws are loosened and PPF removed, estimated 15-30 minutes.
Percentage of planned mastoidectomy reachable by robot | During the use of the PPF, estimated 15-30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Robert F. Labadie, MD, PhD, Principal Investigator — Vanderbilt University Medical Center; Robert J. Webster, PhD, Study Director — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No